CLINICAL TRIAL: NCT01551719
Title: Clinical Usefulness of Mic/Breakpoint Ratio and Penetration in Tissues. A Prospective Study of Clinical Validation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Guglielmo Borgia, Full Professor, Federico II University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 52/11
Record Dates: First submitted 2012-02-29; First posted 2012-03-13 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Infection of Skin and/or Subcutaneous Tissue
Keywords: Bacterial infection of skin or soft tissues
MeSH Terms: conditions — Cellulitis; Skin Diseases, Bacterial | interventions — Cephalosporins; Linezolid; Vancomycin; Daptomycin; Teicoplanin; Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Procedure (phase I) (No Intervention): Antibiotic prescription following in vitro sensitivity test according to each surgeon's will.
- Implemented procedure (Experimental): Prescription following in vitro sensitivity test implemented with MIC/Breakpoint ratio and penetration of antibiotic in the site of infection, according to each surgeon's will.
  Interventions: Behavioral: Implemented procedure

INTERVENTIONS:
Behavioral: Implemented procedure — Prescription following in vitro sensitivity test implemented with MIC/Breakpoint ratio and penetration of antibiotic in the site of infection.
  Other Names: MIC/Breakpoint ratio and tissue penetration for available antibiotics e.g.; - Semisynthetic Penicillins; - Cephalosporins; - Linezolid; - Vancomycin; - Daptomycin; - Teicoplanin; - Tigecycline
  Arms: Implemented procedure

SUMMARY:
The general objective of the study is to assess whether the implementation of the antibiotic essay with the Breakpoint/MIC ratio and data on penetration of the antibiotic in the site of infection may improve the outcome of infections compared to using only the standard procedures.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Bacterial infections, with microbiological isolation, in one of the following tissues: skin, soft tissue or surgical wound infections

Exclusion Criteria:

* Age < 18 years
* Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Complete recovery rate from infection | At the end of treatment (an expected average of 10 days)
  Complete resolution of fever, leukocytosis, and any local signs of infection

SECONDARY OUTCOMES:
Time to recovery from infection. | At the end of treatment (an expected average of 10 days)
  Days to recovery completely from infection.
Partial response | At the end of treatment (an expected average of 10 days)
  Improvement of fever, leukocytosis, and any local signs of infection
Rate of non responders | At the end of treatment (an expected average of 10 days)
  Treatment failure, relapse and death. Failure is defined as no improvement or even worsening of the signs and symptoms of infection.
  Relapse is defined as the resumption of infection with the same organism at any body part within one month after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Borgia, Principal Investigator — Federico II University
Locations (2):
- Italy (2):
  - University of Naples Federico II, Naples, Naples
  - University of Naples Federico II, Naples